CLINICAL TRIAL: NCT05131386
Title: Phase II Multicohort Trial of Trabectedin and Low-dose Radiation Therapy in Advanced/Metastatic Sarcomas
Brief Title: Multicohort Trial of Trabectedin and Low-dose Radiation Therapy in Advanced/Metastatic Sarcomas
Acronym: SYNERGIAS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo Espanol de Investigacion en Sarcomas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEIS-75
Record Dates: First submitted 2021-11-11; First posted 2021-11-23 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Soft Tissue Sarcoma; Bone Tumors; Small Round-cell Sarcomas
Keywords: Osteosarcoma; Chondrosarcoma; Ewing's sarcoma; Rhabdomyosarcoma; Desmoplastic small round-cell tumors
MeSH Terms: conditions — Sarcoma; Bone Neoplasms; Osteosarcoma; Chondrosarcoma; Sarcoma, Ewing; Rhabdomyosarcoma | interventions — Trabectedin

STUDY DESIGN:
Intervention Model Description: Phase II, multicohort, single arm, open-label, multicenter, international clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multicohort trial of trabectedin and low-dose radiation therapy in advanced/metastatic sarcomas (Experimental): Premedication
  4 mg oral dexamethasone 24h and 12h before trabectedin administration, 20 mg IV dexamethasone 30 minutes before treatment. Ondansetron or analogue will also be given prior to trabectedin.
  Medication
  Trabectedin at 1.5 mg/m2 24-h IV CI along with radiation therapy (30 Gy, 3 Gy/day for 10 days for non-extremity location and 45 Gy, 1.8 Gy/day for 25 days for extremity location of target lesion(s)), starting within 1 hour after the first trabectedin infusion withdrawal (day 2)) will be given every 3 weeks up to progression or intolerance.
  Interventions: Drug: Trabectedin

INTERVENTIONS:
Drug: Trabectedin — ET-743, Yondelis (vials of 1 mg). Route of administration: intravenous infusion
  Other Names: Yondelis

SUMMARY:
Phase II, multicohort, single arm, open-label, multicenter, international clinical trial with three cohorts (cohort A: Soft tissue sarcoma, cohort B: Bone tumors (osteosarcoma, chondrosarcoma and cohort C: Small round-cell sarcomas (Ewing's sarcoma, rhabdomyosarcoma, desmoplastic small round-cell tumors and other small round cell sarcomas)) with 7 sites in Spain.

Main objective: To evaluate the overall response rate (ORR) in the irradiated nodules according to RECIST v1.1 criteria.

Treatment

Medication

Trabectedin at 1.5 mg/m2 24-h IV CI along with radiation therapy (30 Gy, 3 Gy/day for 10 days for non-extremity location and 45 Gy, 1.8 Gy/day for 25 days for extremity location of target lesion(s)), starting within 1 hour after the first trabectedin infusion withdrawal (day 2)) will be given every 3 weeks up to progression or intolerance.

Premedication

4 mg oral dexamethasone 24h and 12h before trabectedin administration, 20 mg IV dexamethasone 30 minutes before treatment. Ondansetron or analogue will also be given prior to trabectedin.

DETAILED DESCRIPTION:
Cohort A: Soft tissue sarcomas (2nd or further line): A proportion of 10% of ORR will be considered as not promising, whereas an ORR of 35% will be considered promising in this population. With a type I error α of 0.05 and a power of 0.90, 27 patients were estimated in this cohort. With Simon's two-stage optimal design,36 at least 2 responses have to be obtained over the 11 first patients. Then, additional 16 eligible patients will be accrued up to 27 patients. If at least 6 patients show response, further investigation of this scheme is warranted.

Cohort B: Bone tumors (osteosarcoma, chondrosarcoma) (2nd or further line): A proportion of 3% of ORR will be considered as not promising, whereas an ORR of 20% will be considered promising in this population. With a type I error α of 0.05 and a power of 0.90, 29 patients were estimated in this cohort. With Simon's two-stage optimal design,36 at least 1 response has to be obtained over the 12 first patients. Then, additional 17 eligible patients will be accrued up to 29 patients. If at least 3 patients show response, further investigation of this scheme is warranted.

Cohort C: Small round-cell sarcomas (Ewing's sarcoma, rhabdomyosarcoma, desmoplastic small round-cell tumors and other small round-cell sarcomas) (3rd or further line): A proportion of 15% of ORR will be considered as not promising, whereas an ORR of 40% will be considered promising in this population. With a type I error α of 0.05 and a power of 0.90, 29 patients were estimated in this cohort. With Simon's two-stage optimal design,36 at least 3 response has to be obtained over the 13 first patients. Then, additional 16 eligible patients will be accrued up to 29 patients. If at least 8 patients show response, further investigation of this scheme is warranted.

Taking into account that 10% of enrolled patients might not be evaluable (losses), an extra amount of 3 patients may be recruited per cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must provide written informed consent prior to performance of study-specific procedures and must be willing to comply with treatment and follow up. Informed consent must be obtained prior to start of the screening process. Procedures conducted as part of the patient's routine clinical management (e.g. blood count, imaging tests, etc.) and obtained prior to signature of informed consent may be used for screening or baseline purposes as long as these procedures are conducted as specified in the protocol.
2. Age: 16-75 years.
3. Patients must have a diagnosis of soft tissue sarcoma (cohort A), bone tumors (osteosarcoma, chondrosarcoma) (cohort B) or small round-cell sarcomas (Ewing's sarcoma, rhabdomyosarcoma, desmoplastic small round-cell tumors and other small round cell sarcomas) (cohort C), with metastasis or locally advanced disease, and not suitable for metastasectomy or surgical resection or not oncologically recommended metastasectomy. A centralized diagnosis will be performed, and the central diagnosis confirmation will be mandatory prior to enrollment (tumor sample must be available and sent during screening).
4. Disease distribution allows meeting with normal tissue constraints of radiation therapy. Radiation oncologist must confirm this point, taking into account that the dose for extremities will be 45 Gy while for non-extremity will be 30 Gy.
5. Those lesions considered for radiation therapy must be related with a clinically relevant symptom. It is not necessary to irradiate all the lesions within one organ. Irradiating pulmonary lesions with infiltration of pleural serosa should be discouraged.
6. Patients must have documentation of disease progression within 6 months prior to study entry.
7. The patient must have been considered eligible for systemic chemotherapy. Patients should had received at least one line of systemic therapy (anthracycline-based in the case of Cohort A-STS, unless the patient is not candidate for treatment with anthracyclines), with a maximum of three previous lines for advanced/metastatic disease are allowed as long as trabectedin has not been included.
8. The following sarcoma types are eligible:

   * Soft tissue sarcoma
   * Bone tumors (osteosarcoma, chondrosarcoma)
   * Small round-cell sarcomas (Ewing's sarcoma, rhabdomyosarcoma, desmoplastic small round-cell tumors and other small round cell sarcomas)
9. Measurable disease, according to RECIST v1.1 criteria.
10. Performance status ≤ 1 (ECOG).
11. Adequate respiratory functions: FEV1 > 1L; DLCO > 40% (patients with pulmonary target lesions).
12. Adequate bone marrow function (hemoglobin ≥ 9 g/dL, leukocytes ≥ 3,000/mm3, absolute neutrophil count (ANC) ≥ 1,500/mm3, platelets ≥ 100,000/mm3). Patients with creatinine clearance (based on Cockroft and Gault) ≥30 ml/min, albumin ≥ 25 g/L, ALT and AST ≤ 2.5 times the ULN, total bilirubin ≤ ULN, CPK ≤ 2.5 times ULN, alkaline phosphatase ≤ 2.5 times the ULN are acceptable. If the increase of alkaline phosphatase is > 2.5 times the ULN, then the alkaline phosphatase liver fraction and/or GGT must be ≤ ULN.
13. Men or women of childbearing potential must use an effective method of contraception before entry into the study and throughout the trial treatment and for 6 months after the last dose of trabectedin. Women of childbearing potential must have a negative urine pregnancy test before study entry.
14. Normal cardiac function with a LVEF ≥ 50% by echocardiogram or MUGA.
15. HBV and HCV serologies must be performed prior to enrollment. If HbsAg is positive it is recommended to reject the existence of replicative phase (HbaAg+, DNA VHB+). If these were positives the inclusion is not recommended, remaining at investigators' discretion the preventive treatment with lamivudine. If a potential patient is positive for anti-HCV antibodies, presence of the virus should be ruled out with a qualitative PCR, or the patient should NOT be included in the study (if a qualitative PCR cannot be performed then patient will not be able to enter the study)
16. Patient must have a central venous catheter for treatment, required for trabectedin administration.

Exclusion Criteria:

1. Previous treatment with trabectedin or previous treatment with radiotherapy (this latter just in case the previous radiotherapy treatment does not allow the radiotherapy treatment of this study due to tissue constrains).
2. Liver inclusion in irradiation fields is not permitted, not even partially.
3. Normal tissue constrains for radiation therapy.
4. Performance status ≥ 2 (ECOG).
5. Plasma bilirubin > ULN.
6. Creatinine clearance <30ml/min.
7. History of other neoplastic disease with the exception of basal cell carcinoma or in situ cervical cancer adequately treated or no evidence of recurrence for more than 5 years after primary tumor treatment.
8. Severe chronic obstructive pulmonary disease (COPD) or other severe pulmonary diseases.
9. Significant cardiovascular disease (for example, dyspnea > 2 NYHA).
10. Significant systemic diseases grade 3 or higher on the NCI-CTCAE v5.0 scale, that limit patient availability, or according to investigator judgment may contribute significantly to treatment toxicity.
11. Uncontrolled bacterial, mycotic or viral infections.
12. Known positive test for infection by human immunodeficiency virus (HIV).
13. Women who are pregnant or breast-feeding.
14. Psychological, familiar, social or geographic circumstances that limit the patient's ability to comply with the protocol or informed consent.
15. Patients who have participated in another clinical trial and/or have received any other investigational product in the last 30 days prior to enrollment.
16. Histologies other than those described in inclusion criteria.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2021-05-28 (Actual); Primary Completion 2024-07-28 (Estimated); Study Completion 2024-07-28 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) in the irradiated nodules | 6 weeks
  ORR is defined as the number of subjects with a best overall response (BOR) of complete response (CR) or partial response (PR) only in the irradiated nodules divided by the number of response evaluable subjects (according to RECIST v1.1 criteria and based on central radiology review). This is considered a good surrogate for palliative relief.

SECONDARY OUTCOMES:
Overall response rate (ORR) considering all the lesions | 6 weeks
  ORR is defined as the number of subjects with a best overall response (BOR) of complete response (CR) or partial response (PR) considering all the lesions divided by the number of response evaluable subjects (according to RECIST v1.1 criteria and based on central radiology review).
Progression-free survival rate (PFSR) at 6 months considering all the lesions | 6 months
  Efficacy measured by the PFSR at 6 months according to RECIST v1.1 criteria based on central radiology review. PFSR at 6 months is defined as the percentage of patients who did not experience progression (considering all the lesions) or death due to any cause since the date of enrollment until month 6 after date of enrollment.
Median progression-free survival (mPFS) | 6 months
  Efficacy measured by the mPFS according to RECIST v1.1 criteria based on central radiology review. mPFS is defined as the median of time in months between the date of enrollment and the date of progression (considering all the lesions) or death due to any cause.
Time to progression (TTP) of irradiated nodules | 6 weeks
  TTP is defined as the time in months between the date of enrollment and the date of progression of irradiated nodules (not including deaths) (according to RECIST v1.1 criteria and based on central radiology review).
Overall survival (OS) | 6 months
  OS is defined as the time in months between the date of enrollment and the date of death due to any cause. OS will be censored on the last date a subject was known to be alive.
Variations in pain using the Brief Pain Inventory - Short Form (BPI-SF) | 3 weeks
  Variations from baseline will be assessed on day 1 of every cycle (before trabectedin administration) until cycle 10 and then on day 1 every other cycle (cycle 12 day 1, cycle 14 day 1…).
Variations in quality of life using the QLQ-C30 EORTC v3.0 questionnaire. | 3 weeks
  Variations in quality of life will be assessed at baseline (within 7 days with respect to enrollment), on day 1 of every cycle (before trabectedin administration) until cycle 10 and then on day 1 every other cycle (cycle 12 day 1, cycle 14 day 1…).
Safety profile measured by adverse event type, incidence, severity, time of appearance, and related causes | 3 years
  Toxicity will be assessed through physical explorations and laboratory tests. Toxicity will be graded and tabulated by using CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Andrés Redondo, Principal Investigator — Hospital Universitario La Paz; Claudia Valverde, Principal Investigator — Hospital Universitari Vall d'Hebrón; Katarina Majercakova, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Josefina Cruz, Principal Investigator — Hospital Universitario de Canarias; Rosa Álvarez, Principal Investigator — Hospital General Universitario Gregorio Marañón; Antonio Casado, Principal Investigator — Hospital San Carlos, Madrid; Javier Martín Broto, Study Director — Hospital Universitario Fundación Jiménez Díaz
Locations (7):
- Spain (7):
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - Hospital Universitari Vall d'Hebrón, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No